CLINICAL TRIAL: NCT06406335
Title: Impact of A Multidimensional Health Education Program on Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: ADHD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rasha Saad, Assistant professor of Epidemiology, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Health Education Program ADHD
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: ADHD
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: To measure the impact of a multidimensional health education program on patients' adherence to the healthy life style and behavioral therapy , and to correlate it with severity of ADHD symptoms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- An intervention study (a quasi-experimental design) (Other): a quasi-experimental design pre &post
  Interventions: Other: Health education program

INTERVENTIONS:
Other: Health education program — Impact of A Multidimensional Health Education Program on Attention deficit hyperactivity disorder (ADHD)

SUMMARY:
To measure the impact of a multidimensional health education program on patients' adherence to the healthy life style and behavioral therapy , and to correlate it with severity of ADHD symptoms

DETAILED DESCRIPTION:
Attention-deficit/hyperactivity disorder (ADHD) is a chronic neurodevelopmental disorder whose etiology is the result of complex interactions between multiple factors, including genetic, biological, and environmental influences. Attention deficit hyperactivity disorder (ADHD) is a condition that affects people's behavior. People with ADHD can seem restless, may have trouble concentrating, and may act on impulse. Symptoms of ADHD tend to be noticed at an early age and may become more noticeable when a child's circumstances change, such as when they start school. Most cases are diagnosed when children are 3 to 7 years old, but sometimes it's diagnosed later in childhood .

A mean worldwide prevalence of attention-deficit hyperactivity disorder (ADHD), or hyperkinetic disorder (HKD), of ~2.2% overall (range, 0.1-8.1%) has been estimated in children and adolescents (aged <18 years) . Regarding the prevalence of ADHD in Arabic countries, results from previous studies showed that it reached 9.4-21.8% in Egypt ,and 11.6% in Saudi Arabia .

Several harmful consequences are associated with ADHD, including deficient academic/work performance, social isolation, aggressive behavior (including delinquency and illegal acts), and even premature death from unnatural causes (such as accidents) Undesirable lifestyle factors could contribute directly to inattention and/or hyperactivity symptoms, numerous mechanisms exist that could mediate such effects, such as secondary effects on energy level, immune function, and epigenetic change.

Study findings showed that children with ADHD were approximately two times as likely to have a healthy lifestyle index that is lower than children without ADHD Multiple studies on alternative interventions for ADHD aim at the prevention of ADHD progression and targeting the underlying triggers (such as stress, poor sleep, overstimulation, technology or dietary plans). On the basis that making adequate lifestyle changes to minimize these triggers could contribute to better control of ADHD symptoms .

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with mild and moderate ADHD not receiving medications or behavioral therapy, aged 6-9 years, and parents are motivated to participate in the lifestyle modification program.

Exclusion Criteria:

* Children with severe form of ADHD or with comorbid psychiatric disorders rather than disruptive behavior disorders, and children with an intelligence quotient score below 80 were excluded.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
change in Conners' Parent Rating Scale-Revised, Long Version (CPRS-R-L) | 6 months
  change in mean score Conners' Parent Rating Scale-Revised, Long Version (CPRS-R-L). the Conners' Parents Rating Scale consists of eighty items that need to be rated from zero to 3 (zero means no, 3 means very frequent. the Conners' Rating Scales use the T-score standardized measure to assess results. If a child's T-score is less than 60, that means they don't have ADHD. If the child has a T-score that's higher than 60, that means they likely have ADHD. If the score is higher than 70, their ADHD symptoms are severe)

SECONDARY OUTCOMES:
change in BMI after intervention | 6 months
  change in the mean of BMI after intervention

CONTACTS AND LOCATIONS:
Overall Officials: rasha saad Hussein, MD, Principal Investigator — Faculty of medicine Ain shams univrsity
Locations (1):
- faculty of medicine Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No